CLINICAL TRIAL: NCT05621382
Title: A Comparison of Radiographic and Visual Analysis Methods for Determining Pelvic Misalignments.
Status: Completed | Type: Observational
Sponsor: Sherman College of Straight Chiropractic (Other)
Responsible Party: Principal Investigator, Daniel J. Becker, D.C., Assistant Professor, Sherman College of Straight Chiropractic
Other Study IDs: ShermanCSC
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Gonstead, Chiropractic, Pelvic Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

SUMMARY:
This study looks to compare pelvic misalignments visualized during patient inspection to actual pelvic misalignments derived from x-ray mensuration.

DETAILED DESCRIPTION:
This study looks to compare pelvic misalignments of 30 subjects visualized before x-ray set up to the actual misalignments derived from x-ray mensuration. 30 outpatients at the Sherman College of Chiropractic Health Center were randomly chosen to participate, and were having x-rays taken as part of their normal course of care in order prevent unnecessary radiation exposure. Patients were told to march in place as they were positioned to the x-ray bucky. Once the patient was set to the bucky, the bucky was moved out of the way and the patient was visualized by a health center intern. The intern evaluated gluteal widths, gluteal fold heights, and foot flare. The bucky was then replaced without patient movement and x-rays were then taken. Two doctors with experience in Gonstead line analysis for the pelvis who were blinded to the x-ray findings, measured pelvic misalignments and the results were compared to the visual analysis.

ELIGIBILITY:
Receiving x-rays as part of their normal course of care at the Sherman College of Chiropractic Health Center - There were no exclusion criteria

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients who presented at a chiropractic college health center who were receiving x-rays as part of their care plan.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
A Comparison of Radiographic and Visual Analysis Methods for Determining Pelvic Misalignments. | 7 months
  visual analysis of the pelvis should correlate to radiographic mensuration

CONTACTS AND LOCATIONS:
Locations (1):
- Sherman College of Chiropractic, Spartanburg, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No